CLINICAL TRIAL: NCT04592380
Title: A Randomized Parallel Group Controlled Comparison Study of Clevidipine Versus Placebo or Standard of Care for Dyspnea and Blood Pressure Control in Acute Heart Failure (PRONTO II)
Brief Title: Clevidipine vs Placebo or Standard of Care for Dyspnea and Blood Pressure Control in AHF
Acronym: PRONTO II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Product was divested to Chiesi USA, who decided to not move forward with study.
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-CLV-13-03; PRONTO II (Other: The Medicines Company (Sponsor))
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dyspnea; Hypertension; Acute Heart Failure
MeSH Terms: conditions — Dyspnea; Hypertension | interventions — Double-Blind Method; clevidipine; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stage 1: Clevidipine (double-blinded) (Experimental): Clevidipine (0.5 mg/mL in 20% lipid emulsion) will be administered in a double-blinded fashion intravenously to all patients randomized to the clevidipine arm in Stage 1. Clevidipine will be initiated at an initial rate of 2 mg/h for the first 1.5 minutes (90 seconds) and titrated thereafter per the Food and Drug Administration (FDA) approved clevidipine label, to achieve the target SBP +/- 5 mmHg. If the target SBP is achieved at any of the titration doses, that rate may be continued for up to 24 hours. If the desired BP lowering effect is not attained within 30 minutes or not maintained thereafter, any alternative antihypertensive agent may be used per institutional treatment practice, with or without stopping the study drug infusion.
  Interventions: Drug: Stage 1: Clevidipine (double-blinded)
- Stage 1: Placebo (double-blinded) (Placebo Comparator): Placebo will be administered in a double-blinded fashion intravenously to all patients randomized to the clevidipine arm in Stage 1. Placebo will be initiated at an initial rate of 2 mg/h for the first 1.5 minutes (90 seconds) and titrated thereafter according to the same dosing instructions as for clevidipine to achieve the target SBP +/- 5 mmHg. If the target SBP is achieved at any of the titration doses, that rate may be continued for up to 24 hours. If the desired BP lowering effect is not attained within 30 minutes or not maintained thereafter, any alternative antihypertensive agent may be used per institutional treatment practice, with or without stopping the study drug infusion.
  Interventions: Drug: Stage 1: Placebo (double-blinded)
- Stage 2: Clevidipine (open-label) (Experimental): Clevidipine (0.5 mg/mL in 20% lipid emulsion) will be administered in an open-label fashion intravenously to all patients randomized to the clevidipine arm in Stage 2, following the same dosing instructions as in the clevidipine arm in Stage 1. If the desired BP lowering effect is not attained within 30 minutes or not maintained thereafter, any alternative antihypertensive agent may be used per institutional treatment practice, with or without stopping the study drug infusion.
  Interventions: Drug: Stage 2: Clevidipine (open-label)
- Stage 2: Standard of Care (open-label) (Active Comparator): For patients randomized to SOC, the infusion must be continuous, administered per the institution's treatment practice, and dose titration must be performed to a maximum allowed or maximum tolerated dose to achieve target SBP. If treatment with an alternative IV anti-hypertensive agent is required, the patient will be transitioned to an alternative IV antihypertensive agent according to the institutional standard of care.
  Interventions: Drug: Stage 2: Standard of Care (open-label)

INTERVENTIONS:
Drug: Stage 1: Clevidipine (double-blinded) — Patients may be transitioned to an oral antihypertensive medication as necessary. When such a transition is required, then approximately 1 hour prior to the anticipated cessation of the double-blinded clevidipine infusion, an oral antihypertensive agent may be administered. The clevidipine infusion may be down-titrated or terminated at any time following administration of the oral agent, in order to achieve the desired BP level.
  Other Names: Cleviprex; clevidipine
  Arms: Stage 1: Clevidipine (double-blinded)
Drug: Stage 1: Placebo (double-blinded) — Patients may be transitioned to an oral antihypertensive medication as necessary. When such a transition is required, then approximately 1 hour prior to the anticipated cessation of the double-blinded placebo infusion, an oral antihypertensive agent may be administered. The placebo infusion may be down-titrated or terminated at any time following administration of the oral agent, in order to achieve the desired BP level.
  Other Names: Intralipid
  Arms: Stage 1: Placebo (double-blinded)
Drug: Stage 2: Clevidipine (open-label) — Patients may be transitioned to an oral antihypertensive medication as necessary. When such a transition is required, then approximately 1 hour prior to the anticipated cessation of the clevidipine infusion, an oral antihypertensive agent may be administered. The clevidipine infusion may be down-titrated or terminated at any time following administration of the oral agent, in order to achieve the desired BP level.
  Other Names: Cleviprex; clevidipine
  Arms: Stage 2: Clevidipine (open-label)
Drug: Stage 2: Standard of Care (open-label) — Transition to oral antihypertensive medication from SOC IV antihypertensive is per institutional practice.
  Arms: Stage 2: Standard of Care (open-label)

SUMMARY:
The purpose of this study is to evaluate dyspnea improvement and other parameters of efficacy and safety in acute heart failure (AHF) patients receiving an intravenous (IV) infusion of clevidipine in comparison to standard of care (SOC) and placebo.

DETAILED DESCRIPTION:
Randomization will occur in two stages. Stage 1 patients will be randomized in a double-blinded manner in a 1:1 ratio to receive either clevidipine or placebo IV infusion. Upon completion of Stage 1, Stage 2 patients will be randomized in an open-label manner in a 1:1 ratio to receive either clevidipine or standard of care (SOC) IV infusion. At the time of randomization, a patient-specific, prespecified systolic blood pressure (SBP) target range will be determined and recorded prior to study drug treatment. Up to 500 patients may be enrolled to achieve a total of 100 Stage 1 and 300 Stage 2 patients with confirmed AHF per protocol.

A Data Safety Monitoring Board will be utilized periodically throughout the study to monitor the safety of patients. Adverse events will be assessed for 7 days post-study randomization or hospital discharge, whichever occurred sooner. Serious adverse events (SAEs) were assessed for 30 days following study randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and providing
* Presentation consistent with AHF as manifest by pulmonary congestion
* Dyspnea score (sitting) ≥ 50 mm on a 100 mm visual analog scale
* In Stage 1, baseline SBP ≥130 - 160 mmHg (measured immediately prior to initiation of study drug); in Stage 2, baseline SBP ≥ 130 mmHg

Exclusion Criteria:

* Administration of an IV or oral antihypertensive agent within the previous 2 hours of randomization (short acting oral or sublingual nitrates are permitted)
* Chest pain and/or electrocardiogram (ECG) with ST segment changes consistent with acute coronary syndrome
* Known or suspected aortic dissection
* Acute myocardial infarction (AMI) within the prior 14 days
* Dialysis-dependent renal failure
* Requirement for immediate endotracheal intubation
* Suspected pregnancy or breast feeding female
* Intolerance or allergy to calcium channel blockers
* Allergy to soybean oil or lecithin
* Known liver failure, cirrhosis or pancreatitis
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change in dyspnea VAS score from baseline at 3 hours post-baseline | Immediately prior to study drug administration (baseline) to 3 hours post-baseline

SECONDARY OUTCOMES:
Median time to reach target BP within the first 30 minutes | Study drug initiation through the first 30 minutes of study drug infusion
Percentage of patients who require rescue therapy (ie, receive any alternative IV antihypertensive drug) within the first 30 minutes | Study drug initiation through the first 30 minutes of study drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: William F Peacock, MD, FACEP, Principal Investigator — Baylor College of Medicine
Locations (9):
- United States (9):
  - Drug Research and Analysis Corporation/Jackson Hospital, Montgomery, Alabama
  - University of Arizona Medical Center, Tucson, Arizona
  - Washington University School of Medicine, St Louis, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Stony Brook University and Medical Center, Stony Brook, New York
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas